CLINICAL TRIAL: NCT01161485
Title: Reduction of Drug Use and HIV Risk Among Out-of-Treatment Methamphetamine Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 10-0518
Record Dates: First submitted 2010-07-09; First posted 2010-07-13 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: HIV Infections
Keywords: HIV Infections; Treatment; Methamphetamine
MeSH Terms: conditions — HIV Infections | interventions — HIV Testing; Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HIV Testing and Counseling (Active Comparator): HIV Testing and Counseling
  Interventions: Behavioral: HIV Testing and Counseling
- Contingency Management (CM) (Active Comparator): Contingency management is based on Skinner's principles of operant conditioning in behavioral psychology, dating back to the 1930s (Skinner 1938). The basis of this model is that behavior is learned and reinforced by environmental contingencies that reward or punish.
  Interventions: Behavioral: HIV Testing and Counseling; Behavioral: Contingency Management
- CM with Strengths-based case management (Experimental): Strengths-based case management (SBCM) is a specific type of case management that is based on the following principles: 1) clients are most successful when they identify and use their strengths, abilities, and assets; 2) goal-setting is guided by the clients' perceptions of their own needs; 3) the client-case manager relationship is promoted as essential; 4) a creative approach to the use of the community will lead to the discovery of needed resources; and 5) case management is conducted in the community.
  Interventions: Behavioral: HIV Testing and Counseling; Behavioral: Contingency Management; Behavioral: Strengths-based case management

INTERVENTIONS:
Behavioral: HIV Testing and Counseling — A manualized individual-level model consisting of two education and counseling sessions that structurally bracket confidential HIV antibody screening.
Behavioral: Contingency Management — In voucher-based CM programs, drug users who submit urine samples that are negative for specified drugs are reinforced with vouchers. Based on operant conditioning, CM rewards those who comply with the targeted behavior and does not reward when compliance is not achieved. In this study a mid-value reinforcement CM schedule will be used in order to balance community cost concerns with the need to show comparative efficacy in reducing meth use and concomitant sex risk behaviors in a largely unstudied risk group. Participants in the CM arm will be asked to come to the study site three times a week to leave a urine sample, get the result, and will then be offered a voucher if their urine is clean and given brief verbal feedback.
  Arms: CM with Strengths-based case management; Contingency Management (CM)
Behavioral: Strengths-based case management — Strengths-based case management (SBCM) is a specific type of case management that is based on the following principles: 1) clients are most successful when they identify and use their strengths, abilities, and assets; 2) goal-setting is guided by the clients' perceptions of their own needs; 3) the client-case manager relationship is promoted as essential; 4) a creative approach to the use of the community will lead to the discovery of needed resources; and 5) case management is conducted in the community. It differs from more traditional case management models that emphasize resource brokerage and client advocacy in its recognition that only the individual can change his/her behavior.
  Arms: CM with Strengths-based case management

SUMMARY:
There is a need to identify and test effective strategies to reduce meth use and human immunodeficiency virus (HIV) risk behaviors in heterosexuals. This project will compare the efficacy of a manually-driven HIV testing and counseling (HIV T/C) intervention, with HIV T/C plus a manualized Contingency Management (CM), with HIV T/C plus CM plus a manualized Strengths-Based Case Management (CM/SBCM) model. As HIV T/C is the standard of care, the investigators are testing to determine if the investigators can enhance this standard. The specific aims and hypotheses of this protocol are:

1. To compare the relative efficacy of HIV T/C vs. CM vs. CM/SBCM on reducing drug use, specifically meth use. Hypothesis 1: CM/SBCM will reduce drug use more than those in CM (which will have more reduction than HIV T/C), potentially mediated through increased service utilization.
2. To compare the relative efficacy of HIV T/C vs. CM vs. CM/SBCM on reducing HIV and STI risk behaviors, specifically sex risk behaviors but also needle risk for injection drug users (IDUs). Hypothesis 2: CM/SBCM will have greater decreases in HIV risk behaviors than those in CM (which will have greater decreases than HIV T/C), potentially mediated through reduced drug use.
3. To compare the relative efficacy of HIV T/C vs. CM vs. CM/SBCM on improving mental health status. Hypothesis 3: CM/SBCM will have greater improvements in mental health status than those in CM (which will have greater improvements than HIV T/C), potentially mediated through increased service utilization and reduction of drug use, and potentially moderated by baseline meth use.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Be competent (not too intoxicated or mentally disabled) to give informed consent at the time of the interview
* Meth use (verified through urine drug screening and a self-report of meth use of at least 4 times per month for the last 3 months)
* Self-reported sex with someone of the opposite sex in last 30 days
* Ability to provide a reliable address and phone number for contact
* Not in drug treatment in the past 30 days
* Willingness to be tested for HIV at baseline and follow-up
* Not transient and no know reason why he/she will not be available for follow-up interviews
* Not currently mandated by the criminal justice system to receive treatment based on self-report.

Exclusion Criteria:

* Participation in drug treatment in the past 30 days
* Currently participating in another Project Safe study
* Pregnant or attempting to become pregnant
* Intoxicated or impaired mentally to the point that they cannot voluntarily consent to participate tin the project and/or respond to the interview

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 502 (Actual)
Dates: Start 2010-08; Primary Completion 2015-06-13 (Actual); Study Completion 2016-05-25 (Actual)

PRIMARY OUTCOMES:
Reduction of drug use, specifically methamphetamine | 12-month follow-up interview
Reduction of HIV and STI risk behaviors, specifically sex risk behaviors but also needle risk for injection drug users | 12-month follow-up interview
Improved mental health status | 12-month follow-up interview

CONTACTS AND LOCATIONS:
Overall Officials: Karen F Corsi, ScD, MPH, Principal Investigator — University of Colorado, Denver
Locations (1):
- Project Safe, Denver, Colorado, United States